CLINICAL TRIAL: NCT07392879
Title: Bringing the Outdoors In: Virtual Nature Walks for Depression in Multiple Sclerosis (MS) Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Apple Inc. (Industry); The International Organization of Multiple Sclerosis Nurses Inc (Unknown)
Responsible Party: Principal Investigator, Hala Darwish, Associate Professor of Nursing, University of Michigan
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HUM00267042
Record Dates: First submitted 2026-01-29; First posted 2026-02-06 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Progressive Multiple Sclerosis; Depression
Keywords: Immersive virtual reality (VR)
MeSH Terms: conditions — Multiple Sclerosis, Chronic Progressive; Depression | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: There are 3 groups (2 groups that take standard care (SC) treatment for depression will be randomized) that participants are assigned to: 1) VR plus SC therapy followed by washout and SC only; 2) SC for 8 weeks washout then VR plus SC. The third group will be VR only (not on any treatment for depression and not randomized).
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Virtual reality plus standard care (SC) then SC alone - randomized group (Experimental): Participants in this group are maintained on antidepressants or psychotherapy and will receive VR nature sessions alongside participants' current depression treatments. This will be followed by a 1-week washout period, after which they crossover to standard care only.
  Interventions: Device: Virtual Reality; Other: Standard care
- Standard care alone then Virtual reality plus SC- randomized group (Experimental): Participants in this group are maintained on standard depression treatments and will continue standard care for eight weeks. This will be followed by a 1-week washout period and crossover to VR plus Standard Care.
  Interventions: Device: Virtual Reality; Other: Standard care
- Virtual Reality - non-randomized group (Experimental): Participants that are not receiving any treatment for depression will receive VR nature sessions for 8 weeks without depression treatments for eight weeks followed by 1 week washout and 8 weeks of no VR.
  Interventions: Device: Virtual Reality

INTERVENTIONS:
Device: Virtual Reality — Participant will have 8 weeks of immersive VR nature-based experiences. Participants are expected to use the VR headset three times per week. Headsets will contain a prototype application (app) developed by Explore POV. This app will include approximately one hour of footage showcasing 15-25 different nature experiences, that will shuffle every time participants access it. Participants will have the option to choose between 5, 10, or 15 minutes, sessions while answering weekly surveys regarding their experiences.
Other: Standard care — Participants that are in the randomized groups will continue on antidepressants or psychotherapy during the study per their standard care. Participants in the non-randomized group don't receive any treatment for their depression and will continue not to receive anything for this during the study.
  Arms: Standard care alone then Virtual reality plus SC- randomized group; Virtual reality plus standard care (SC) then SC alone - randomized group

SUMMARY:
This trial explores the use of immersive virtual reality (VR) nature-based experiences as a supplementary treatment for depression in individuals with progressive multiple sclerosis (MS). This study will evaluate the feasibility and efficacy of at-home VR deployment using the Apple Vision Pro, an advanced device that offers enhanced resolution, immersion, and usability compared to earlier VR systems.

The study hypotheses include:

* The integration of VR nature-based experiences with standard care will be feasible, acceptable, and will result in greater reductions in depressive symptoms compared to standard care or VR-only interventions.
* The integration of VR nature-based experiences with standard care will result in greater reductions in stress and anxiety, better sleep, less insomnia, and improved fatigue compared to standard care alone or VR-only interventions.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of progressive Multiple Sclerosis (MS, primary or secondary) by a neurologist or an MS center
* Patient-Reported Outcomes Measurement Information System (PROMIS) Depression T-scores >55 at baseline
* Ability to provide informed consent and participate in VR sessions at home
* For Some Participants (Groups 1 and 2) currently receiving antidepressant or psychotherapy treatments (Selective Serotonin Reuptake Inhibitors (SSRIs), Serotonin-Norepinephrine Reuptake Inhibitors (SNRIs), or psychotherapy) for the management of depression

Exclusion Criteria:

* Severe cognitive impairments or visual deficits that may interfere with VR use, including contraindications like agoraphobia, claustrophobia, or motion sickness
* Current participation in other clinical trials targeting depression
* Severe psychiatric conditions that require hospitalization, or suicidal ideation, passive or active, psychosis, or active substance and alcohol abuse (score greater than 1 on CAGE (Cut down, Annoyed, Guilty, Eye-opener) Adapted to Include Drugs (CAGE-AID))
* Another neurological or autoimmune disease per protocol
* Participants that require vision correction, unless that vision correction is mild (± 1), or the participant has prescription contact lenses.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-15 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Changes to the Patient-Reported Outcomes Measurement Information System (PROMIS) Depression short form 8b scores | Baseline, 9-10 weeks and 20-21 weeks
  This is an 8-item evaluating various aspects of depression, including negative mood, anhedonia, feelings of worthlessness, and cognitive impairments. Each item is rated on a 5-point Likert scale ranging from never (1) - always (5). Scores range from 8-40 with a higher score indicating greater symptom severity.
Virtual Reality (VR) Sessions completed over 8 weeks | 8-week VR intervention
  A benchmark of 70% will indicate adequate feasibility and acceptability.
Qualitative feedback on the VR Neuroscience Questionnaire during the intervention (groups 1 and 3) | 1-8 weeks (during VR)
  The modified scale for this project uses 10 questions that participants will answer about the VR experience, rated from 1 (extremely low or extremely difficult) to 7 (extremely high or extremely easy). The scores range from 10 to 70, with higher scores indicating greater experience. A benchmark of 70% indicates adequate feasibility and acceptability, with participant satisfaction ratings above 80%.
Qualitative feedback with Semi-structured interviews for participants that received VR | Weeks 9-10, Weeks 20- 21
  Semi-structured interviews with 20 random participants (6-7 from each group) who received the VR treatment to capture participants' subjective experiences at the midpoint and end of the intervention.
  The interview questions will focus on emotional changes, engagement levels, and feedback on the intervention's implementation.
Enrollment rate | Recruitment period (2 years)
  Feasibility will be assessed via enrollment. Recruitment will be quantified by enrollment rates relative to the number of eligibility screenings.
Retention rates | Baseline - 21 weeks
  Feasibility: Retention will be evaluated through the percentage of participants who complete the entire study duration, targeting a benchmark of at least 70%.
Adherence to VR intervention | 8-week VR intervention
  Feasibility: Adherence to 5-15-minute sessions 3 times per week over 8 weeks
Dropout reasons | Baseline - 21 weeks
Hardware/software issues | During 8 weeks of VR

SECONDARY OUTCOMES:
Change to the PROMIS Anxiety short form scores of the VR experience | Baseline, 8 weeks (after VR)
  This consists of eight items assessing various dimensions of anxiety, including feelings of fear, worry, hyperarousal, and somatic symptoms. Each item is rated on a 5-point Likert scale ranging from never (1) - always (5). Scores range from 8-40 with a higher score indicating greater anxiety.
Change to the patient perceived stress scale (PSS-10) | Baseline, 8 weeks (after VR)
  It comprises 10 items that assess how unpredictable, uncontrollable, and overloaded respondents find their lives. Each item is rated on a 5-point Likert scale ranging from Never (0) to Very Often (4).
  The total score ranges from 0 to 40, with higher scores indicating greater perceived stress. While there are no established cut-off scores, higher scores suggest higher levels of perceived stress.
Change in Sleep based on the Pittsburgh Sleep Quality Index (PSQI) | Baseline, 8 weeks (after VR)
  It comprises 19 items, generating seven component scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication, and daytime dysfunction. Each component is scored from 0 to 3, with higher scores indicating greater dysfunction. The component scores are summed to yield a global PSQI score ranging from 0 to 21. A global score greater than 5 suggests poor sleep quality.
Change in the Insomnia Severity Index (ISI) | Baseline, 8 weeks (after VR)
  This is a brief self-report tool that evaluates the nature, severity, and impact of insomnia. It consists of seven items, each rated on a 5-point Likert scale (0 = no problem to 4 = very severe problem), assessing areas such as difficulty falling asleep, staying asleep, satisfaction with sleep, and the extent to which sleep problems interfere with daily functioning. The total score ranges from 0 to 28, with higher scores indicating more severe insomnia. Interpretation of scores is as follows: 0-7 (no clinically significant insomnia), 8-14 (subthreshold insomnia), 15-21 (moderate insomnia), and 22-28 (severe insomnia).
Change in the PROMIS Fatigue | Baseline, 8 weeks (after VR)
  The PROMIS Fatigue Short Form 7a is a validated self-report instrument designed to assess fatigue over the past seven days. It consists of seven items that evaluate the frequency and severity of fatigue and its impact on daily activities. Each item is rated on a 5-point Likert scale ranging from "Never" (1) to "Always" (5). The raw scores are summed and converted into standardized T-scores, with a mean of 50 and a standard deviation of 10, based on the U.S. general population. Higher T-scores indicate greater fatigue severity. A change of 3 to 5 T-score points is generally considered clinically meaningful.

CONTACTS AND LOCATIONS:
Overall Officials: Hala Darwish, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No